CLINICAL TRIAL: NCT00896337
Title: A Boston Scientific Trial of the EPIC™ Nitinol Stent System in the Treatment of Atherosclerotic Lesions in Iliac Arteries
Brief Title: EPIC Nitinol Stent System in the Treatment of Atherosclerotic Lesions in Iliac Arteries
Acronym: ORION
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2020
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Results first posted 2012-07-03 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-04

CONDITIONS: Iliac Artery Stenosis
Keywords: iliac artery stenosis; claudication; atherosclerotic iliac disease; peripheral vascular disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases | interventions — Dual Anti-Platelet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ORION (Experimental): All subjects who meet the inclusion criteria and are enrolled in this trial will be treated with iliac artery stenting with the Epic™ Nitinol Stent System.
  Interventions: Device: Epic™ Nitinol Stent System; Drug: Anti-platelet therapy; Drug: Anti-coagulation therapy

INTERVENTIONS:
Device: Epic™ Nitinol Stent System — The Epic™ Nitinol Stent System is comprised of two components: the implantable nitinol endoprosthesis and the stent delivery system.
Drug: Anti-platelet therapy — Investigators must prescribe concomitant anti-platelet medication consistent with current clinical practice. Anti-platelet therapy should be administered preprocedure and continued throughout participation in the trial.
Drug: Anti-coagulation therapy — Anti-coagulation therapy must be administered during the procedure consistent with current clinical practice.

SUMMARY:
The ORION study is being conducted to determine whether the Epic™ Nitinol Stent for primary stenting of iliac atherosclerotic lesions shows acceptable performance at 9 months.

DETAILED DESCRIPTION:
ORION is a prospective, single arm, non-randomized, multicenter study. A subject could receive a maximum of 2 study stents for up to 2 target lesions. A maximum of 1 non-target lesion in 1 non-target vessel could be treated with a commercially approved treatment during the index procedure.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic, symptomatic iliac artery atherosclerotic disease (Rutherford/Becker category 1, 2, 3 or 4)
* Lifestyle-limiting claudication or rest pain
* De novo or restenotic lesions in the common and/or external iliac artery
* Subjects with bilateral disease may have only one target lesion treated per side
* Two target lesions may be treated with a maximum of two stents (if two target lesions are treated, each lesion must be covered with a maximum of one stent)
* Length of diseased segment(s) <=13 cm and treatment is planned with no more than 2 overlapped Epic™ stents
* Baseline diameter stenosis >= 50% (operator visual assessment)
* Reference vessel diameter >= 5 mm and <=11 mm
* At least one sufficient ipsilateral infrapopliteal run-off vessel
* Origin of profunda femoris artery is patent

Exclusion Criteria:

* Target vessel with in-stent restenosis
* Acute critical limb ischemia
* Tissue loss (Rutherford/Becker category 5 or 6)
* Any major amputations to the target limb
* Any minor amputation of the target limb in the last 12 months. If a minor amputation occurred greater than 12 months, stump needs to be completely healed.
* Life expectancy less than 24 months due to other medical co-morbid condition(s) that could limit the subject's ability to participate in the trial, limit the subject's compliance with the follow-up requirements, or impact the scientific integrity of the trial
* Known hypersensitivity or contraindication to contrast dye that, in the opinion of the investigator, cannot be adequately pre-medicated.
* Intolerance to antiplatelet, anticoagulant, or thrombolytic medications
* Platelet count < 150,000 mm3 or > 600,000 mm3
* Serum creatinine > 2.0 mg/dL
* Dialysis-dependent end stage renal disease
* Pregnancy
* Current participation in another drug or device trial that has not completed the primary endpoint or that may potentially confound the results of this trial
* Known allergy to Nitinol
* Presence of arterial lesions (with the exception of renal, carotid or short, focal SFA lesions) requiring intervention within 30 days of the index procedure - Superficial femoral artery occlusion in the limb supplied by target vessel
* Heavily calcified and/or excessively tortuous lesions in the target vessel as determined by angiography
* Target lesion is within or near an aneurysm
* Persistent, intraluminal thrombus of the proposed target lesion post-thrombolytic therapy
* Perforated vessel as evidenced by extravasation of contrast media
* Vascular graft, aneurysm or postsurgical stenosis of the target vessel
* Multiple lesions in the same target vessel unable to be treated with a maximum of two stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-05; Primary Completion 2011-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela G. Grady, Ph.D., Study Director — Boston Scientific Corporation; Daniel G Clair, MD, Principal Investigator — The Cleveland Clinic
Locations (28):
- United States (28):
  - St. Joseph's Hospital, Tucson, Arizona
  - Brandon Regional Hospital, Brandon, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mediquest Research at Munroe Regional Medical Center, Ocala, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Parkview Hospital-Parkview Research Center, Fort Wayne, Indiana
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Trinity Terrace Park, Davenport, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - North Memorial Medical Center, Robbinsdale, Minnesota
  - Mount Sinai Medical Center, New York, New York
  - Mid-Carolina Cardiology - Presbyterian Hospital, Charlotte, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - MeritCare Hospital, Fargo, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - University of Oklahoma Health Science Center, Oklahoma City, Oklahoma
  - UPMC - Shadyside Hospital, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Erlanger Medical Center, Chattanooga, Tennessee
  - St. Thomas Research Institute, Nashville, Tennessee
  - VA North Texas Health Care System, Dallas, Texas
  - Baptist Hospital of San Antonio, San Antonio, Texas
  - Fletcher Allen Health Care, Burlington, Vermont

REFERENCES:
- [Derived] Clair DG, Adams J, Reen B, Feldman R, Starr J, Diaz-Cartelle J, Dawkins KD. The EPIC nitinol stent system in the treatment of iliac artery lesions: one-year results from the ORION clinical trial. J Endovasc Ther. 2014 Apr;21(2):213-22. doi: 10.1583/13-4560.1. PMID 24754280

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of up to 133 subjects was planned; 125 subjects were enrolled at 28 centers in the United States from May 14, 2009 to December 14, 2010.
Period: Overall Study
Arm/Group | ORION
Started | 125
Completed | 100
Not Completed | 25
Not completed — Death | 7
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Arm/Group | ORION
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 80
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 81
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 3
  Caucasian | 112
  Black of African heritage | 8
  American Indian or Alaska Native | 1
  Asian | 0
  Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 125
General Medical History [Number; unit: Participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    Smoking, Ever | 121
    Medically Treated Diabetes | 42
    Hyperlipidemia Requiring Medication | 98
    Hypertension Requiring Medication | 95
    History of Chronic Obstructive Pulmonary Disease | 31
Cardiac History [Number; unit: Participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    History of Coronary Artery Disease | 73
    History of Myocardial Infarction | 36
    History of Congestive Heart Failure | 10
    Stable Angina | 15
    Unstable Angina | 1
    Silent Ischemia | 0
    Previous Percutaneous Coronary Intervention | 46
    Previous Coronary Artery Bypass Graft | 22
Peripheral Vascular History [Number; unit: Participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participants
    History of Peripheral Vascular Surgery | 10
    History of Other Peripheral Endovascular Intervent | 25
    History of Claudication | 116
Neurologic/Renal History [Number; unit: participants] — The same participant may be included in more than one category or not all participants may contribute to a category, therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  participants
    History of Transient Ischemic Attack | 5
    History of Cerebrovascular Accident | 7
    History of Renal Insufficiency | 9
    History of Renal Percutaneous Intervention | 6
Lesion Characteristic: Target Lesion Vessel [Number; unit: Lesions] — These data are reported per lesion. A participant could have more than one lesion, therefore, the number of lesions reported for this baseline measure does not equal the total number of participants in the group.
  Lesions
    Left Common Iliac Artery | 58
    Left External Iliac Artery | 16
    Right Common Iliac Artery | 58
    Right External Iliac Artery | 28
Lesion Characteristic: Lesion Location [Number; unit: Lesions] — These data are reported per lesion. A participant could have more than one lesion, therefore, the number of lesions reported for this baseline measure does not equal the total number of participants in the group.
  Lesions
    Ostial | 100
    Proximal | 35
    Mid | 12
    Distal | 13
Lesion Characteristics: Size [Mean (Standard Deviation); unit: millimeters] — These data are reported per lesion.
  millimeters
    Reference Vessel Diameter | 7.69 (1.79)
    Minimum Lumen Diameter | 2.20 (1.34)
    Lesion Length | 31.04 (22.13)
Lesion Characteristic: Diameter Stenosis [Mean (Standard Deviation); unit: percent] — These data are reported per lesion. A participant could have more than one lesion, therefore, the number of lesions reported for this baseline measure does not equal the total number of participants in the group.
  percent | 71.51 (16.27)
Lesion Characteristics [Number; unit: Lesions] — These data are reported per lesion. A participant could have more than one lesion; therefore, the number of lesions reported for this baseline measure does not equal the total number of participants in the group. The same participant's lesion may also be included in more than one category or not all participants may contribute to a category.
  Lesions
    Concentric Lesion | 72
    Eccentric Lesion | 88
    > 45 Degree Bend | 1
    > 90 Degree Bend | 0
    Thrombus | 0
    Calcification, Non/Mild | 37
    Calcification, Moderate | 45
    Calcification, Severe | 78
    Ulcerated | 29
    Total Occlusion | 26
    Aneurysm | 10

OUTCOME MEASURES:

1. Primary Outcome: Device- and/or Procedure-related Major Adverse Events (MAE)
Description: MAE is defined as any device-related or index procedure-related death within 30 days, myocardial infarction during index hospitalization, target vessel revascularization through 9 months, or amputation of the index limb through 9 months
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 7 participants were not evaluable.
Measure: Number; unit: percentage of participants
Groups:
- Epic Stent: Participants treated with iliac artery stenting using the Epic™ Nitinol Stent System.
Arm/Group | Epic Stent
Number analyzed (Participants) | 118
percentage of participants | 3.4
Statistical Analysis 1: Comparison: Epic Stent; MAE rate was compared to a predefined performance goal of 17.0%, based on literature-derived expected rate of 8.0% for iliac stenting plus a 9.0% margin. Study had 87% statistical power to show the MAE rate (accounting for 9-month attrition of <=15%) is less than the performance goal, assuming a 9-month MAE rate of 8.0%. If the exact one-sided 95% upper confidence bound of the observed rate is lower than the performance goal, the Epic stent would be considered to have acceptable performance; Test type: Superiority or Other; p < 0.0001, One-sided exact-test — A one-sided exact-test was used to test the hypothesis that the primary endpoint rate in the Epic-treated cohort is less than the predefined performance goal of 17.0%; 9-month major adverse event rate = 3.4, 95% CI 2-sided [0.9 to 8.5]

2. Secondary Outcome: Death
Description: Death is classified as follows. Cardiac death: death due to immediate cardiac cause, death of unknown cause is classified as cardiac death, including all procedure related deaths including those related to concomitant treatment; Vascular death: death due to cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause; Non-cardiovascular death: any death not covered by the above definitions
Time Frame: 30 Days
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 4 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 121
percentage of participants | 0.0

3. Secondary Outcome: Death
Description: Death is classified as follows. Cardiac death: death due to immediate cardiac cause; death of unknown cause is classified as cardiac death, including all procedure related deaths including those related to concomitant treatment; Vascular death: death due to cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause; Non-cardiovascular death: any death not covered by the above definitions
Time Frame: 9 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Epic Stent: Subjects treated with iliac artery stenting using the Epic™ Nitinol Stent System.
Arm/Group | Epic Stent
Number analyzed (Participants) | 118
percentage of participants | 0.8

4. Secondary Outcome: Death
Description: as for outcome 3
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 11 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 114
percentage of participants | 1.8

5. Secondary Outcome: Death
Description: as for outcome 3
Time Frame: 2 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 17 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 108
percentage of participants | 3.7

6. Secondary Outcome: Death
Description: as for outcome 3
Time Frame: 3 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 18 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 107
percentage of participants | 6.5

7. Secondary Outcome: Amputation of Index Limb
Description: Major amputation: amputation of the lower limb at the ankle level or above Minor amputation: amputation of forefoot or toes
Time Frame: 9 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 118
percentage of participants | 0.0

8. Secondary Outcome: Amputation of Index Limb
Description: as for outcome 7
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 13 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 112
percentage of participants | 0

9. Secondary Outcome: Amputation of Index Limb
Description: as for outcome 7
Time Frame: 2 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 19 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 106
percentage of participants | 0

10. Secondary Outcome: Amputation of Index Limb
Description: as for outcome 7
Time Frame: 3 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 25 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 100
percentage of participants | 0

11. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: Target vessel revascularization (TVR) is defined as any surgical or percutaneous intervention to the target vessel(s) after the index procedure. A TVR is considered ischemia-driven if the culprit lesion stenosis is ≥50% by quantitative angiography and the subject has ischemic symptoms.
  A TVR is considered ischemia-driven if the culprit lesion diameter stenosis is ≥70% even in the absence of clinical or functional ischemia.
Time Frame: 30 Days
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 121
percentage of participants | 2.5

12. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 11
Time Frame: 9 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 118
percentage of participants | 3.4

13. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 11
Time Frame: 1 Year
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 112
percentage of participants | 3.6

14. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 11
Time Frame: 2 Years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 106
percentage of participants | 8.5

15. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 11
Time Frame: 3 Years
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 24 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 101
percentage of participants | 12.9

16. Secondary Outcome: Myocardial Infarction (MI)
Description: Definition of myocardial infarction: New Q-waves in ≥2 leads lasting ≥0.04 sec with creatine kinase- myoglobin band (CK-MB)/troponin above upper limit of normal (ULN); if no new Q-waves elevation of post-procedure CK levels >2.0× ULN with positive CK-MB, or, if the assay for CK-MB was not performed, elevation of CK levels >2.0× ULN with positive troponin. Drawing a CK-MB or troponin is mandated if CK is greater than 2× ULN. If no CK-MB or troponin was drawn, CK >2× ULN will be considered an MI. ULN is determined per local laboratory specifications.
Time Frame: Index hospitalization
Population: Analysis was intention to treat; all participants in the study were evaluated to provide the information needed for this endpoint
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 125
percentage of participants | 0.0

17. Secondary Outcome: Technical Success
Description: Residual lesion stenosis <=30% based on visual assessment immediately postprocedure
Time Frame: Index procedure
Population: as for outcome 16
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Groups:
- Epis Stent: Participants treated with iliac artery stenting using the Epic™ Nitinol Stent System
Arm/Group | Epis Stent
Number analyzed (Participants) | 125
Number analyzed (Lesions) | 166
percentage of lesions | 100

18. Secondary Outcome: Procedure Success
Description: Technical success (residual lesion stenosis <=30% based on visual assessment immediately postprocedure) and no in-hospital major adverse events (device- or index procedure-related death, myocardial infarction, target vessel revascularization or amputation of the index limb).
Time Frame: In hospital (1-2 days post procedure)
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 125
percentage of participants | 99.2

19. Secondary Outcome: Early Clinical Success
Description: Improvement in Rutherford classification by 1 class as compared to baseline. Rutherford Classification is used to assess lower extremity ischemia as shown below:
  Class 0 = Asymptomatic Class 1 = Mild claudication Class 2 = Moderate claudication Class 3 = Severe claudication Class 4 = Ischemic rest pain Class 5 = Minor tissue loss - non-healing ulcer, focal gangrene with diffuse pedal edema
Time Frame: Hospital Discharge
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 12 participants were not evaluable
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 113
percentage of participants | 44.2

20. Secondary Outcome: Early Clinical Success
Description: as for outcome 19
Time Frame: 30 Days
Population: as for outcome 19
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 113
percentage of participants | 87.6

21. Secondary Outcome: Late Clinical Success
Description: as for outcome 19
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint. There were 16 participants not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Epic Stent
Number analyzed (Participants) | 109
percentage of patients | 89.9

22. Secondary Outcome: Late Clinical Success
Description: as for outcome 19
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint. There were 19 participants not evaluable.
Measure: Number; unit: percentage of patients
Arm/Group | Epic Stent
Number analyzed (Participants) | 106
percentage of patients | 95.3

23. Secondary Outcome: Early Hemodynamic Success
Description: Improvement in ankle-brachial index (ABI) by ≥0.1 from the pre-procedure value and not deteriorated by >0.15 from the maximum post-procedure value. Reported per limb.
Time Frame: Hospital Discharge
Population: as for outcome 19
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 113
Number analyzed (Limbs) | 152
percentage of limbs | 61.2

24. Secondary Outcome: Early Hemodynamic Success
Description: as for outcome 23
Time Frame: 30 Days
Population: as for outcome 19
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 113
Number analyzed (Limbs) | 151
percentage of limbs | 66.2

25. Secondary Outcome: Late Hemodynamic Success
Description: as for outcome 23
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 8 participants were not evaluable.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 117
Number analyzed (Limbs) | 141
percentage of limbs | 66.7

26. Secondary Outcome: Late Hemodynamic Success
Description: as for outcome 23
Time Frame: 1 Year
Population: as for outcome 4
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 114
Number analyzed (Limbs) | 132
percentage of limbs | 63.6

27. Secondary Outcome: Rutherford Classification Distribution
Description: Rutherford Classification is used to assess lower extremity ischemia as shown below:
  0 = Asymptomatic
  1. = Mild claudication
  2. = Moderate claudication
  3. = Severe claudication
  4. = Ischemic rest pain
  5. = Minor tissue loss - non-healing ulcer, focal gangrene with diffuse pedal edema
Time Frame: Pre-procedure/baseline
Population: as for outcome 16
Measure: Number; unit: percentage of participants
Groups:
- Epic Stent: Participants who received the Epic Stent during the index procedure.
Arm/Group | Epic Stent
Number analyzed (Participants) | 125
percentage of participants
  Asymptomatic | 0.0
  Mild Claudication | 7.2
  Moderate Claudication | 33.6
  Severe Claudication | 54.4
  Ischemic Rest Pain | 4.8
  Minor Tissue Loss | 0.0
  Major Tissue Loss | 0.0

28. Secondary Outcome: Rutherford Classification Distribution
Description: as for outcome 27
Time Frame: Post-procedure
Population: Analysis was intention to treat; all participants in the study were evaluated to provide the information needed for this endpoint; 12 participants were not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 113
percentage of participants
  Asymptomatic | 17.7
  Mild Claudication | 20.4
  Moderate Claudication | 35.4
  Severe Claudication | 23.0
  Ischemic Rest Pain | 3.5
  Minor Tissue Loss | 0
  Major Tissue Loss | 0

29. Secondary Outcome: Rutherford Classification Distribution
Description: as for outcome 27
Time Frame: 30 Days
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 113
percentage of participants
  Asymptomatic | 65.6
  Mild Claudication | 16.8
  Moderate Claudication | 13.3
  Severe Claudication | 4.4
  Ischemic Rest Pain | 0
  Minor Tissue Loss | 0
  Major Tissue Loss | 0

30. Secondary Outcome: Rutherford Classification Distribution
Description: Rutherford Classification is used to assess lower extremity ischemia as shown below:
  Class 0 = Asymptomatic Class 1 = Mild claudication Class 2 = Moderate claudication Class 3 = Severe claudication Class 4 = Ischemic rest pain Class 5 = Minor tissue loss - non-healing ulcer, focal gangrene with diffuse pedal edema Class 6 = Major tissue loss
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; there were 16 participants not evaluable.
Measure: Number; unit: percentage of participants
Groups:
- Epic Stent: Participants who received the Epic Stent
Arm/Group | Epic Stent
Number analyzed (Participants) | 109
percentage of participants
  Asymptomatic | 63.3
  Mild Claudication | 18.3
  Moderate Claudication | 15.6
  Severe Claudication | 2.8
  Ischemic Rest Pain | 0.0
  Minor Tissue Loss | 0.0
  Major Tissue Loss | 0.0

31. Secondary Outcome: Rutherford Classification Distribution
Description: as for outcome 30
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; there were 19 participants not evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 106
percentage of participants
  Asymptomatic | 76.4
  Mild Claudication | 12.3
  Moderate Claudication | 10.4
  Severe Claudication | 0.9
  Ischemic Rest Pain | 0
  Minor Tissue Loss | 0
  Major Tissue Loss | 0

32. Secondary Outcome: Acute Stent Thrombosis
Description: Angiographic documentation of an acute, complete occlusion of a previously successfully treated lesion and/or Angiographic documentation of a flow-limiting thrombus within, or adjacent to, a previously successfully treated lesion
  Acute stent thrombosis is defined as occurring <=24 hours following the trial procedure. Subacute stent thrombosis is defined as occurring >24 hours to <=30 days following the trial procedure.
Time Frame: 24 Hours
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 121
percentage of participants | 0.0

33. Secondary Outcome: Sub-acute Stent Thrombosis
Description: Angiographic documentation of an acute, complete occlusion of a previously successfully treated lesion and/or Angiographic documentation of a flow-limiting thrombus within, or adjacent to, a previously successfully treated lesion
  Acute stent thrombosis is defined as occurring less than or equal to 24 hours following the trial procedure. Subacute stent thrombosis is defined as occurring >24 hours to less than or equal to 30 days following the trial procedure.
Time Frame: >24 Hours to <=30 Days Post-index procedure
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 121
percentage of participants | 2.5

34. Secondary Outcome: Stent Thrombosis
Description: Angiographic documentation of an acute, complete occlusion of a previously successfully treated lesion and/or Angiographic documentation of a flow-limiting thrombus within, or adjacent to, a previously successfully treated lesion
  Late stent thrombosis is defined as >30 days to 365 days following the trial procedure.
Time Frame: 9 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 118
percentage of participants | 2.5

35. Secondary Outcome: Stent Thrombosis
Description: as for outcome 34
Time Frame: 1 Year
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 112
percentage of participants | 2.7

36. Secondary Outcome: Stent Thrombosis
Description: Angiographic documentation of an acute, complete occlusion of a previously successfully treated lesion and/or Angiographic documentation of a flow-limiting thrombus within, or adjacent to, a previously successfully treated lesion
  Very late stent thrombosis is defined as >365 days following the trial procedure.
Time Frame: 2 Years
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 106
percentage of participants | 2.8

37. Secondary Outcome: Stent Thrombosis
Description: as for outcome 36
Time Frame: 3 Years
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Epic Stent
Number analyzed (Participants) | 101
percentage of participants | 4.0

38. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: Target lesion revascularization (TLR) is any surgical or percutaneous intervention to the target lesion(s) after the index procedure. A TLR will be considered ischemia-driven if the target lesion diameter stenosis is ≥50% by quantitative angiography and the subject has ischemic symptoms. A TLR will be considered ischemia-driven if the lesion diameter stenosis is ≥70% even in the absence of clinical or functional ischemia.
Time Frame: 30 Days
Population: as for outcome 2
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 121
Number analyzed (Lesions) | 161
percentage of lesions | 1.9

39. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 38
Time Frame: 9 Months
Population: as for outcome 1
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 118
Number analyzed (Lesions) | 157
percentage of lesions | 3.2

40. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 38
Time Frame: 1 Year
Population: as for outcome 8
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 112
Number analyzed (Lesions) | 150
percentage of lesions | 3.3

41. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 38
Time Frame: 2 Years
Population: as for outcome 9
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 106
Number analyzed (Lesions) | 143
percentage of lesions | 5.6

42. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 38
Time Frame: 3 Years
Population: as for outcome 15
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 101
Number analyzed (Lesions) | 139
percentage of lesions | 10.1

43. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: Ratio between the systolic pressure measured at the ankle and the systolic pressure measured in the arm as follows:
  Ankle: The systolic pressure will be measured in the index limb at the arteria dorsalis pedis and/or the arteria tibialis posterior. If both pressures are measured, the highest pressures will be used for the ABI calculation.
  Brachial: The systolic pressure will be measured in both arms, and the highest of both pressures will be used for the ABI calculation.
Time Frame: Pre-procedure/baseline
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 125
Number analyzed (Limbs) | 159
ratio | 0.79 (0.18)

44. Secondary Outcome: Ankle-Brachial Index
Description: as for outcome 43
Time Frame: Hospital Discharge (1-2 days post-procedure)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 125
Number analyzed (Limbs) | 155
ratio | 0.96 (0.17)

45. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: as for outcome 43
Time Frame: 30 Days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 121
Number analyzed (Limbs) | 153
ratio | 0.99 (.015)

46. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: as for outcome 43
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 15 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 110
Number analyzed (Limbs) | 142
ratio | 0.97 (0.17)

47. Secondary Outcome: Ankle-Brachial Index (ABI)
Description: as for outcome 43
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 16 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: ratio
Units Other Than Participants: Limbs
Arm/Group | Epic Stent
Number analyzed (Participants) | 109
Number analyzed (Limbs) | 135
ratio | 0.96 (0.17)

48. Secondary Outcome: Primary Patency
Description: Systolic velocity ratio (SVR) is the ratio of the measurement of systolic velocity in 2 arterial regions as determined by duplex ultrasound (DUS). Primary patency (defined per lesion) is defined as DUS SVR ≤2.5 with no target lesion revascularization, bypass of the target lesion, or amputation.
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 30 participants were not evaluable
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 95
Number analyzed (Lesions) | 122
percentage of lesions | 95.9

49. Secondary Outcome: Primary Patency
Description: as for outcome 48
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 50 participants were not evaluable
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 99
percentage of lesions | 93.9

50. Secondary Outcome: Primary-assisted Patency (PAP)
Description: Systolic velocity ratio (SVR) is the ratio of the measurement of systolic velocity in 2 arterial regions as determined by duplex ultrasound (DUS). Primary-assisted patency (defined per lesion) is defined as DUS SVR ≤2.5 with no target lesion revascularization for total occlusion, bypass of the target lesion, or amputation. In 1 subject, SVR was invalid and DUS proximal peak systolic velocity was analyzed to assess restenosis.
Time Frame: 9 Months
Population: as for outcome 48
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 95
Number analyzed (Lesions) | 122
percentage of lesions | 98.4

51. Secondary Outcome: Primary-assisted Patency (PAP)
Description: as for outcome 50
Time Frame: 1 Year
Population: as for outcome 49
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 99
percentage of lesions | 96.0

52. Secondary Outcome: Secondary Patency
Description: Systolic velocity ratio (SVR) is the ratio of the measurement of systolic velocity in 2 arterial regions as determined by duplex ultrasound (DUS). Secondary patency (defined per lesion) is defined as having DUS SVR ≤2.5 in the absence of bypass of the target lesion or amputation. In 1 subject, SVR was invalid and proximal peak systolic velocity was analyzed to assess restenosis.
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to undergo clinical follow up to provide the information needed for this endpoint; 31 participants were not evaluable
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 94
Number analyzed (Lesions) | 120
percentage of lesions | 100

53. Secondary Outcome: Secondary Patency
Description: as for outcome 52
Time Frame: 1 Year
Population: as for outcome 49
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 98
percentage of lesions | 98.0

54. Secondary Outcome: Restenosis Assessed by Duplex Ultrasound
Description: Systolic velocity ratio (SVR) is the ratio of the measurement of systolic velocity in 2 arterial regions as determined by duplex ultrasound (DUS). Restenosis (defined per lesion)is defined as DUS SVR >2.5 or the presence of a target lesion revascularization prior to the DUS examination, regardless of the SVR value. In 1 subject, SVR was invalid and proximal peak systolic velocity by DUS was analyzed to assess restenosis.
Time Frame: 9 Months
Population: as for outcome 48
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 95
Number analyzed (Lesions) | 122
percentage of lesions | 2.5

55. Secondary Outcome: Restenosis Assessed by Duplex Ultrasound
Description: as for outcome 54
Time Frame: 1 Year
Population: as for outcome 49
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Epic Stent
Number analyzed (Participants) | 75
Number analyzed (Lesions) | 99
percentage of lesions | 6.1

56. Secondary Outcome: Walking Impairment Questionnaire Score - Distance
Description: The Walking Impairment Questionnaire is a functional-assessment questionnaire that evaluates walking ability with regard to speed, distance and stair climbing ability as well as the reasons that walking ability might be limited. Range of scores is between 0% and 100% with 100% being the best and 0% being the worst score.
Time Frame: Pre-procedure/baseline
Population: Analysis was intention to treat; all participants in the study were to be evaluated to provide the information needed for this endpoint; one participant was not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 124
units on a scale | 14.56 (19.36)

57. Secondary Outcome: Walking Impairment Questionnaire Score - Distance
Description: as for outcome 56
Time Frame: 9 Months
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 110
units on a scale | 56.35 (38.97)

58. Secondary Outcome: Walking Impairment Questionnaire Score - Distance
Description: as for outcome 56
Time Frame: 1 Year
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 109
units on a scale | 55.88 (38.02)

59. Secondary Outcome: Walking Impairment Questionnaire Score - Speed
Description: as for outcome 56
Time Frame: Pre-procedure/baseline
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 124
units on a scale | 18.38 (19.18)

60. Secondary Outcome: Walking Impairment Questionnaire Score - Speed
Description: as for outcome 56
Time Frame: 9 Months
Population: as for outcome 46
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 110
units on a scale | 48.45 (31.50)

61. Secondary Outcome: Walking Impairment Questionnaire Score - Speed
Description: as for outcome 56
Time Frame: 1 Year
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 109
units on a scale | 47.96 (31.80)

62. Secondary Outcome: Walking Impairment Questionnaire Score-Stair Climbing
Description: as for outcome 56
Time Frame: Pre-procedure/baseline
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 124
units on a scale | 26.14 (26.91)

63. Secondary Outcome: Walking Impairment Questionnaire Score - Stair Climbing
Description: as for outcome 56
Time Frame: 9 Months
Population: Analysis was intention to treat; all participants in the study were to be evaluated to provide the information needed for this endpoint; 15 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 110
units on a scale | 59.39 (38.08)

64. Secondary Outcome: Walking Impairment Questionnaire Score - Stair Climbing
Description: as for outcome 56
Time Frame: 1 Year
Population: Analysis was intention to treat; all participants in the study were to be evaluated to provide the information needed for this endpoint; 17 participants were not evaluable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Epic Stent
Number analyzed (Participants) | 108
units on a scale | 57.72 (37.17)

ADVERSE EVENTS:
Time Frame: 3 Years
Arm/Group | ORION
Serious Adverse Events (participants affected / at risk) | 77/125
Other Adverse Events (participants affected / at risk) | 63/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORION (N=125)
Anaemia (Blood and lymphatic system disorders) | 1 (3)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1)
Angina Pectoris (Cardiac disorders) | 7 (8)
Angina Unstable (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 7 (10)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Coronary Artery Disease (Cardiac disorders) | 4 (5)
Coronary Artery Stenosis (Cardiac disorders) | 3 (3)
Ischaemic Cardiomyopathy (Cardiac disorders) | 2 (2)
Mitral Valve Stenosis (Cardiac disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 3 (3)
Blindness (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 1 (2)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1)
Catheter Site Haematoma (General disorders) | 1 (1)
Catheter Site Haemorrhage (General disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Non-cardiac Chest Pain (General disorders) | 4 (5)
Oedema Peripheral (General disorders) | 1 (1)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 1 (1)
Abdominal Abscess (Infections and infestations) | 1 (1)
Clostridial Infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 6 (7)
Wound Infection (Infections and infestations) | 1 (1)
Drug Toxicity (Injury, poisoning and procedural complications) | 1 (1)
Stent-graft Malfunction (Injury, poisoning and procedural complications) | 2 (2)
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Blood Creatinine Increased (Investigations) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Recurrent Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid Artery Stenosis (Nervous system disorders) | 4 (5)
Diplegia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 2 (2)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Angiodysplasia (Vascular disorders) | 1 (1)
Arterial Stenosis (Vascular disorders) | 1 (1)
Iliac Artery Thrombosis (Vascular disorders) | 2 (2)
Intermittent Claudication (Vascular disorders) | 5 (7)
Peripheral Artery Dissection (Vascular disorders) | 3 (3)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Vascular Occlusion (Vascular disorders) | 1 (1)
Vessel Perforation (Vascular disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute Myocardial Infarction (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Cardiac Failure Congestive (Cardiac disorders) | 3 (3)
Sinus Arrhythmia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 2 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic Polyp (Gastrointestinal disorders) | 1 (1)
Large Intestine Perforation (Gastrointestinal disorders) | 1 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Bronchiectasis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Septic Shock (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Chemical Eye Injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1)
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant Peritoneal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 3 (3)
Convulsion (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Calculus Ureteric (Renal and urinary disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Renal Artery Stenosis (Renal and urinary disorders) | 2 (2)
Renal Failure Acute (Renal and urinary disorders) | 2 (2)
Renal Mass (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 2 (2)
Femoral Arterial Stenosis (Vascular disorders) | 1 (3)
Hypertension (Vascular disorders) | 2 (2)
Iliac Artery Occlusion (Vascular disorders) | 1 (1)
Iliac Artery Stenosis (Vascular disorders) | 6 (6)
Leriche Syndrome (Vascular disorders) | 1 (1)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 1 (1)
Subclavian Steal Syndrome (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ORION (N=125)
Catheter Site Haematoma (General disorders) | 10 (10)
Back Pain (Musculoskeletal and connective tissue disorders) | 14 (17)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 15 (22)
Angina Pectoris (Cardiac disorders) | 7 (7)
Bronchitis (Infections and infestations) | 7 (8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least 45 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.